CLINICAL TRIAL: NCT01542762
Title: Pot-Cast: Thrombosis Prophylaxis During Plaster Cast Lower Leg Immobilisation: Determining the Balance Between Benefits and Risks
Brief Title: Pot-Cast: Thrombosis Prophylaxis During Plaster Cast Lower Leg Immobilisation
Acronym: Pot-Cast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzanne C. Cannegieter, MD PhD (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, Suzanne C. Cannegieter, MD PhD, Study director, Leiden University
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL35774.058.11; 171102001 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Deep Venous Thrombosis; Pulmonary Embolism
Keywords: Deep venous thrombosis; Pulmonary Embolism; Lower leg Cast immobilization
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Heparin, Low-Molecular-Weight; Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LMWH (Experimental): 750 patients with lower leg cast immobilization will be randomized tot receive treatment with a LMWH.
  Interventions: Drug: LMWH
- No intervention (No Intervention): 750 patients with lower leg cast immobilization will be randomized tot receive no treatment with LMWH.

INTERVENTIONS:
Drug: LMWH — Each hospital will use a LMWH according to their own preferences.
  Prophylactic dosage of LMWH (for example nadroparin 2850 IE s.c.) once daily for the duration of the immobilization (average 6 weeks). If the patient's weight is more than 100kg a double dose of LMWH will be given (in case of Nadroparin 5700 IE s.c. once daily).
  Other Names: Nadroparine; Dalteparine
  Arms: LMWH

SUMMARY:
Currently, guidelines and clinical practice differ considerably with respect to use of anticoagulant treatment during cast immobilization of the lower leg. Trials that have been carried out were aimed at efficacy only, had small sample sizes and therefore mainly used asymptomatic thrombosis as endpoint. From these trials an overall risk benefit-balance could not be established, hence the current controversy. In the proposed study the investigators will use relevant symptomatic endpoints in a large cohort of patients. Furthermore the investigators will follow subjects with an adverse event for a longer period, during which the investigators will assess the long term sequelae of these events. Lastly, the investigators will determine high risk groups that will benefit most from anticoagulant treatment.

Objective: Comparative effectiveness research to determine cost-effectiveness of two existing policies, i.e. treatment with low molecular weight heparin (LMWH) during lower leg plaster cast immobilization following surgical or conservative treatment. In addition the investigators will investigate personalized prophylaxis based on genetic and acquired risk factors.

DETAILED DESCRIPTION:
Background:

Currently, guidelines and clinical practice differ considerably with respect to use of anticoagulant treatment during cast immobilization of the lower leg. Trials that have been carried out were aimed at efficacy only, had small sample sizes and therefore mainly used asymptomatic thrombosis as endpoint. From these trials an overall risk benefit-balance could not be established, hence the current controversy exists. In the proposed study we will use relevant symptomatic endpoints in a large cohort of patients. Furthermore we will follow subjects with an adverse event for a longer period, during which we will assess the long term sequelae of these events. Lastly, we will determine high risk groups that will benefit most from anticoagulant treatment.

Objective:

Comparative effectiveness research to determine cost-effectiveness of an existing healthcare policy, i.e. treatment with low molecular weight heparin (LMWH) during lower leg plaster cast immobilization following surgical or conservative treatment. In addition we will investigate personalized prophylaxis based on genetic and acquired risk factors.

Study Design:

A randomized controlled trial comparing a policy with the anticoagulant LMWH to a policy with no anticoagulant in patients with lower leg cast immobilization.

Determination of genetic and acquired risk factors will be performed at the start of the study. Based on the presence or absence of these factors we will assign a risk profile to each patient

Study Population:

The study population will consist of 1500 patients in need for a plaster cast of the lower leg, e.g. after trauma or overuse injuries of ankle and foot. These patients will be recruited from 5 hospitals in the Leiden/Den Haag region over a two-year inclusion period. All patients over 18 years will be eligible, except patients with a contra-indication or an absolute indication for LMWH use

Intervention:

LMWH (for example nadroparin 2850 IE s.c. once daily, > 100kg 5700IE sc) for the duration of the immobilization (average 6-8 weeks) vs no treatment.

Each hospital will use a LMWH according to their own preference.

Blood taken at the emergency department will be analyzed on common single nucleotide polymorphisms (SNPs) known to strongly affect thrombotic risk; on levels of coagulation factors in plasma (of which high or low levels are known to increase the risk). Patients will also be screened on acquired risk factors for thrombosis through a questionnaire.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

We will compare two standard treatment modes that are currently both used depending on the physician's or hospital's preference. The patients in our trial will be subjected to one of these standard treatments. It is therefore not expected that participation will lead to an increased health risk. LMWHs like Nadroparin and Dalteparin are no experimental pharmaceuticals; both have been registered in the Netherlands for these indications since 1989.

Not participating in the trial may, depending on the physician, still lead to treatment with an LMWH.

All patients will need to undergo one venepuncture for blood sampling for the study. This blood sample will be taken at the first day of immobilization. No extra hospital visits are required. Patients will be contacted by an electronic questionnaire 3 weeks and 7 weeks after the start of immobilization and by telephone after three months.

One questionnaire concerning risk factors for thrombosis, bleeding and patients demographics will be filled in at the first day of cast immobilization.

Only subjects with clinically relevant adverse events (and a similar random sample of subjects without a clinically relevant adverse event) will be monitored for a two year period after the event (in total expected to be about 30 subjects). After six months, one year and two years after the event, patients will be seen for clinical examination and quality of life assessment by means of a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

All patients in need of immobilization of the lower leg with a plaster cast (or equivalent of a cast) for a minimum of one week for the following indications:

* Trauma of the lower leg
* Surgery of the lower leg followed by lower leg immobilization with a plaster cast
* Non-traumatic indications

Exclusion Criteria:

* Contra-indications for LMWH use (recent major bleeding, bleeding disorder, allergy)
* Pregnancy
* Pre-existent indication for anticoagulation therapy, either LMWH or vitamin K antagonists.
* History of venous thromboembolism (indication for anticoagulation therapy for prophylaxis of recurrence)
* Mental of physical disability to fulfill study requirements
* Insufficient knowledge of the Dutch language
* Previous participation in the Pot-(K)Cast study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2012-03; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Symptomatic deep venous thrombosis (DVT) | 3 Months
  Symptomatic deep venous thrombosis confirmed with compression ultrasonography
Pulmonary Embolism (PE) | 3 months
  Fatal or non-fatal pulmonary embolism confirmed with:
  * an intraluminal filling defect in segmental or more proximal branches on spiral CT scan, or
  * a perfusion defect of at least 75% of a segment with a local normal ventilation result (high-probability) on ventilation/perfusion lung scan, or
  * detected at autopsy
Major Bleeding | 3 months
  Major bleeding, defined as:
  * a fatal bleeding, or
  * symptomatic bleeding in a critical area or organ, or
  * extrasurgical site bleeding causing a fall in hemoglobin level of 1.24mmol/L (2.0g/dL) or more, leading to transfusion of one or more units of whole blood or red cells, or
  * surgical site bleeding that requires a second intervention or a hemarthrosis interfering with rehabilitation, or surgical site bleeding that needs blood suppletion.

SECONDARY OUTCOMES:
Other clinically relevant bleeding | 3 months
  Other clinically relevant bleeding, defined as overt bleeding not meeting the criteria for major bleeding but associated with medical intervention, unscheduled contact with a physician, (temporary) cessation of study treatment, or associated with discomfort such as pain, or impairment of activities of daily life.
Surgical site infection | 3 months
  Superficial incisional surgical site infection, deep incisional surgical site infection of organ/space surgical site infection according to the definitions of the CDC.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C Cannegieter, PhD, MD, Study Director — Leiden University Medical Center; Rob GHH Nelissen, PhD, MD, Principal Investigator — Leiden University Medical Center
Locations (8):
- Netherlands (8):
  - De Isala Klinieken, Zwolle, Overijssel
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - Groene Hart Ziekenhuis, Gouda, South Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Rijnland Ziekenhuis, Leiderdorp, South Holland
  - Medisch Centrum Haaglanden, The Hague, South Holland
  - HagaZiekenhuis, The Hague, South Holland
  - Bronovo Ziekenhuis, The Hague, South Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Adrichem RA, Nemeth B, Algra A, le Cessie S, Rosendaal FR, Schipper IB, Nelissen RGHH, Cannegieter SC; POT-KAST and POT-CAST Group. Thromboprophylaxis after Knee Arthroscopy and Lower-Leg Casting. N Engl J Med. 2017 Feb 9;376(6):515-525. doi: 10.1056/NEJMoa1613303. Epub 2016 Dec 3. PMID 27959702